CLINICAL TRIAL: NCT02478619
Title: Effects of Preoperative Inspiratory Muscle Training in Patients Undergoing Gastroplasty
Brief Title: Preoperative Inspiratory Muscle Training in Gastroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ada Clarice Gastaldi, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USP 2015-2
Record Dates: First submitted 2015-06-16; First posted 2015-06-23 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2015-06

CONDITIONS: Obesity
Keywords: Obesity; Respiratory Muscle Training; Bariatric Surgery; Breathing exercises; Gastroplasty
MeSH Terms: conditions — Obesity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMT group (Active Comparator): The volunteers will do the respiratory muscle training through a linear inspiratory pressure resistance device (POWERbreathe®) at 50% of the maximal inspiratory pressure.
  Interventions: Other: IMT group
- Control group (Placebo Comparator): Patients will do a placebo respiratory muscle training through a load pressure resistance device (POWERbreathe®) with the minimum load available (10cmH20).
  Interventions: Other: Control group

INTERVENTIONS:
Other: IMT group — Patients will be instructed to do a daily inspiratory muscle training at home with the preset load at 50% of the maximal inspiratory pressure, during 30 minutes for 4 weeks before bariatric surgery.
  They will also receive the routine physical therapy in the post operative period.
  Other Names: Respiratory resistance device (POWERbreathe®)
  Arms: IMT group
Other: Control group — Patients will be instructed to do a daily inspiratory muscle training at home with the minimal inspiratory load of the respiratory resistance device, during 30 minutes for 4 weeks before bariatric surgery. They will also receive the routine physical therapy in the post operative period.
  Arms: Control group

SUMMARY:
The purpose of this study is to assess the effect of preoperative inspiratory muscle training in patients with grade III obesity undergoing bariatric surgery. It will be a double-blind randomized controlled clinical trial with volunteers allocated in two groups that will be compared according to postoperative evolution (pulmonary complications, lung function, strength and endurance of the respiratory muscles and respiratory system resistance).

DETAILED DESCRIPTION:
The prevalence of obesity has a significantly increase in recent years and represents a public health problem due to the increased risk of mortality from various causes. Changes in respiratory system arising from obesity are well established and they include a reduction in compliance with an increased ventilatory work and oxygen consumption with breathing. Bariatric surgery is an alternative surgical treatment of obesity and patients who undergo this surgery are susceptible to post operative pulmonary complications as a result of obesity and also abdominal surgery. The inspiratory muscle training (IMT) used in pre or post operative period can improve muscle strength and endurance, beyond the perception of dyspnea.There are suggestions that the preoperative training may contribute to a best post operative evolution in patients, but these benefits are not clearly defined in the literature. The objective is to evaluate the effects of preoperative IMT in post operative patients undergoing gastroplasty. There will be 40 patients of bariatric surgery group in Ribeirão Preto Medical School of both sexes, BMI>40 kg/m2 and with the appropriate inclusion criteria.They will be assessed by pulmonary function tests, measurement of strength and endurance of respiratory muscles, submaximal exercise tests, dyspnea and quality of life scales. All patients will receive standard treatment and will be randomly divided into two groups, named control group and training group, who will be trained for 4 weeks preoperatively. The patients will be reassessed after 4 weeks of training and on the 15th postoperative return day. The evolution data about pulmonary complications will be collected from the medical records, notes of the medical staff and physical therapy routine service.

ELIGIBILITY:
Inclusion Criteria:

* patients attending the bariatric surgery's ambulatory;
* patients presenting body mass index (BMI) ≥ 40 kg/m2.

Exclusion Criteria:

* acute or chronic pulmonary diseases;
* smoking;
* not stable cardiovascular diseases;
* decompensated diabetes.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Complications | From the first to the 15th post-operative day
  According to Brooks-Brunn (1997) methodology, pulmonary complications will be considered as: cough/sputum production, abnormal breath sounds, temperature ≥ 38°C, chest radiograph documentation of atelectasis or new infiltrate, physician documentation of atelectasis or pneumonia.

SECONDARY OUTCOMES:
Maximal Static Respiratory Pressures | First evaluation: preoperative / before IMT (4 weeks before surgery); Second evaluation: preoperative / after IMT (6-1 days before /surgery); Third evaluation: postoperative / after IMT (15 days after surgery)
  It has beem used a digital manometer (MVD300, Global Med, São Paulo, Brazil) with graduation ranging from 0 to ± 300 cmH2O and adjusted to a rigid mouthpiece, following the proposed model by Black and Hyatt in 1969.
Inspiratory Muscle Endurance Test | First evaluation: preoperative / before IMT (4 weeks before surgery); Second evaluation: preoperative / after IMT (6-1 days before surgery); Third evaluation: postoperative / after IMT (15 days after surgery)
  This measurement is performed by using the POWERbreathe® device at 80% maximal inspiratory pressure, following the ATS/ERS recommendations (2002) and Bellemare & Grassino methodology (1982).
Impulse Oscillometry | First evaluation: preoperative / before IMT (4 weeks before surgery); Second evaluation: preoperative / after IMT (6-1 days before surgery); Third evaluation: postoperative / after IMT (15 days after surgery)
  To perform this measure, it is been used Jaeger® IOS(Jaeger, Wurzburg, Germany) with daily volume and resistance calibration. Data collection happens in different positions: sitting, supine, right lateral decubitus and left lateral decubitus. The parameters are calculated at frequencies between 5 and 35Hz, and will be analyzed the following parameters in this test: resistance (R), reactance (X), reactance area (AX) and resonant frequency (Fres).
Pulmonary Function Test | First evaluation: preoperative / before IMT (4 weeks before surgery); Second evaluation: preoperative / after IMT (6-1 days before surgery); Third evaluation: postoperative / after IMT (15 days after surgery)
  This test is realized by using KoKo Spirometer according ATS/ERS recommendations. The analyzed parameters in this test are: forced vital capacity (FVC), Forced Expiratory Volume in the First Second (FEV1), FEV1/FVC and FEF25-75%.
Six Minute Walking Test | First evaluation: preoperative / before IMT (4 weeks before surgery); Second evaluation: preoperative / after IMT (6-1 days before surgery); Third evaluation: postoperative / after IMT (15 days after surgery)
  Patients walk through a 30-meter corridor faster than they can for 6 minutes, according to ATS considerations. The assessed parameters during this test are: blood pressure, cardiac and respiratory frequencies, peripheral oxygen saturation and Borg's Scale.
Dyspnea's Perception | First evaluation: preoperative / before IMT (4 weeks before surgery); Second evaluation: preoperative / after IMT (6-1 days before surgery); Third evaluation: postoperative / after IMT (15 days after surgery)
  The volunteers answer the mMRC Questionnaire
Life's Quality | First evaluation: preoperative / before IMT (4 weeks before surgery); Second evaluation: preoperative / after IMT (2 days before surgery); Third evaluation: postoperative / after IMT (15 days after surgery)
  The volunteers answer the SF-36 Questionnaire
Level of Physical Activity | First evaluation: preoperative / before IMT (4 weeks before surgery); Second evaluation: preoperative / after IMT (2 days before surgery); Third evaluation: postoperative / after IMT (15 days after surgery)
  The volunteers answer the International Physical Activity Questionnaire (IPAQ).

CONTACTS AND LOCATIONS:
Overall Officials: Ada C Gastaldi, PhD, Principal Investigator — Ribeirão Preto Medicine School - University of São Paulo
Locations (1):
- Ribeirão Preto Medicine School, University of São Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Casali CC, Pereira AP, Martinez JA, de Souza HC, Gastaldi AC. Effects of inspiratory muscle training on muscular and pulmonary function after bariatric surgery in obese patients. Obes Surg. 2011 Sep;21(9):1389-94. doi: 10.1007/s11695-010-0349-y. PMID 21229331
- [Background] Barbalho-Moulim MC, Miguel GP, Forti EM, Campos Fdo A, Costa D. Effects of preoperative inspiratory muscle training in obese women undergoing open bariatric surgery: respiratory muscle strength, lung volumes, and diaphragmatic excursion. Clinics (Sao Paulo). 2011;66(10):1721-7. doi: 10.1590/s1807-59322011001000009. PMID 22012043
- [Background] Kulkarni SR, Fletcher E, McConnell AK, Poskitt KR, Whyman MR. Pre-operative inspiratory muscle training preserves postoperative inspiratory muscle strength following major abdominal surgery - a randomised pilot study. Ann R Coll Surg Engl. 2010 Nov;92(8):700-7. doi: 10.1308/003588410X12771863936648. Epub 2010 Jul 26. PMID 20663275
- [Background] Dronkers J, Veldman A, Hoberg E, van der Waal C, van Meeteren N. Prevention of pulmonary complications after upper abdominal surgery by preoperative intensive inspiratory muscle training: a randomized controlled pilot study. Clin Rehabil. 2008 Feb;22(2):134-42. doi: 10.1177/0269215507081574. Epub 2007 Dec 5. PMID 18057088